CLINICAL TRIAL: NCT02008929
Title: A Single Center, Open-label, Phase II Clinical Trial to Evaluate the Efficacy and Safety of MG4101(Ex Vivo Expanded Allogeneic NK Cell) in Hepatocellular Carcinoma After Curative Resection
Brief Title: to Evaluate the Efficacy and Safety of MG4101(Ex Vivo Expanded Allogeneic NK Cell)
Acronym: MG4101
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, JAE WON JOH, Clinical Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC_ MG4101
Record Dates: First submitted 2013-12-08; First posted 2013-12-11 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: NKCELL
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MG4101 (Other): Ex vivo expanded allogeneic NK cell
  Interventions: Biological: MG4101

INTERVENTIONS:
Biological: MG4101 — Ex vivo expanded allogeneic NK cell
  Other Names: NK cell

SUMMARY:
To see the safety and efficacy of injecting MG4101 as a secondary treatment after curative liver resection on the patient with advanced HCC who has high risk of recurrence.

DETAILED DESCRIPTION:
To see the safety and efficacy of injecting MG4101(Ex vivo expanded allogeneic NK cell) as a secondary treatment after curative liver resection on the patient with advanced HCC who has high risk of recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Under the age of 20 to 69 years of age
2. Child-pugh class A
3. After curative liver resection, diagnosed hepatocellular carcinoma
4. Modified UICC staging : stage 3
5. the women who is childbearing age, agree to maintain adequate contraception measure during clinical trial period.
6. Agreed to participate in this clinical trial, agree to the subject person or legal representative who agrees in writing

Exclusion Criteria:

1. Less than 20 years old, 70 years old or older
2. Metastasis of hepatocellular carcinoma with external parties surgery
3. who had Rupture of hepatocellular carcinoma (HCC)
4. Hepatocellular carcinoma treated with radiofrequency surgery therapeutics (Radiofrequency ablation, RFA), the carotid artery chemical embolization (Transarterial chemoembolization, TACE), underwent radiation therapy, such as topical therapeutics
5. suspected serious infection
6. Who have severe cardiovascular disease (coronary artery disease requiring treatment, heart failure, arrhythmias, myocardial infarction, etc.)
7. Pregnant, planning a pregnancy or breast-feeding women
8. Autoimmune Disease
9. Those who Latest within four weeks of administration of systemic steroids (However, inhalation, intranasal corticosteroids and topical administration of corticosteroids and short-time administration of a blood transfusion, if such reasons are excluded)
10. Latest within four weeks of taking immunosuppressive drugs such as Cyclosporine A
11. Within the last 5 years diagnosed with liver cancer and other malignancies
12. Investigator did not complete or the effectiveness or safety of pharmaceutical products of this clinical trial evaluation for any medical condition that can interfere with characters judged

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Disease free survival, DFS | Disease free survival for 1year
  As of Date for allocation to survival and recurrence of the incident or death from any cause is defined as. 1 year disease-free survival was calculated using Kaplan-Meier estimation and 95% confidence interval and median survival (median survival time) are presented.

SECONDARY OUTCOMES:
Changes in tumor markers | Changes in tumor markers. to be specific, alpha-fetoprotein(AFP), protein induced by vitamin K absence- II(PIVKA-II)
  Basaline(V2) at each visit compared (V6, V8, V9, V10) with respect to variation in average by descriptive statistics (mean, standard deviation, median, minimum, maximum) and presented, in comparison to the group in order Paired t-test or the Wilcoxon's signed rank test for analysis.
Overall survival, OS | Overall survival, OS at the end point of clinical trial
  As of Date for allocation to survival, and the incident was defined as death from any cause.
  1 year overall survival was calculated using Kaplan-Meier estimation and 95% confidence interval and median survival (median survival time) are presented.

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Won Joh, MD., PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kim JM, Cho SY, Rhu J, Jung M, Her JH, Lim O, Choi GS, Shin EC, Hwang YK, Joh JW. Adjuvant therapy using ex vivo-expanded allogenic natural killer cells in hepatectomy patients with hepatitis B virus related solitary hepatocellular carcinoma: MG4101 study. Ann Hepatobiliary Pancreat Surg. 2021 May 31;25(2):206-214. doi: 10.14701/ahbps.2021.25.2.206. PMID 34053923